CLINICAL TRIAL: NCT01147666
Title: A Phase 2, Randomized, Open-Label Active-Comparator (Epoetin Alfa) and Single-Blind Placebo-Controlled, Dose-Ranging Safety and Exploratory Efficacy Study of FG-4592 in Subjects With End-Stage Renal Disease Receiving Maintenance Hemodialysis
Brief Title: Study of Roxadustat (FG-4592) in Participants With End-Stage Renal Disease Receiving Maintenance Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FGCL-4592-040
Record Dates: First submitted 2010-05-20; First posted 2010-06-22 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: End Stage Renal Disease; Anemia
Keywords: Kidney; End Stage Renal Disease; ESRD; Chronic Kidney Disease; CKD; Renal; Anemia; Oral anemia treatment; Hemoglobin levels; Blood count; Erythropoietin; Hemodialysis; Normoresponder; Hyporesponder
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia; Renal Insufficiency, Chronic | interventions — roxadustat; Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Cohort A-1 (Roxadustat 1.0 mg/kg TIW) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 1.0 milligrams (mg)/kg, administered orally 3 times weekly (TIW) in the morning of the day after dialysis (interdialytic days) for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 grams [g]/deciliter [dL]) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-2 (Roxadustat 1.5 mg/kg TIW) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 1.5 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-3 (Roxadustat 2.0 mg/kg TIW) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-4 (Roxadustat 1.8 mg/kg TIW) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 1.8 mg/kg, administered orally TIW for 6 weeks. Participants who have not completed 6-week treatment at the time of Amendment 2, will continue treatment for up to 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-5 (Roxadustat 1.8 mg/kg TIW) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 85-115 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 1.8 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-6 (Roxadustat 1.3 mg/kg TIW) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 1.3 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) will receive tiered, weight-based initial doses of roxadustat (approximately 1.3 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants will receive roxadustat 70 mg, 100 mg, and 150 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) will receive tiered, weight-based initial doses of roxadustat (approximately 1.5 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants will receive roxadustat 70 mg, 120 mg, and 200 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-9 (Roxadustat 2.0 mg/kg) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 85-150 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) (Experimental): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) will receive tiered, weight-based initial doses of roxadustat (approximately 1.5 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants will receive roxadustat 70 mg, 120 mg, and 200 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohorts A (Epoetin Alfa) (Active Comparator): Normoresponsive participants will receive IV epoetin alfa treatments on Day 1, at their prestudy dose and according to their prestudy dosing schedule (TIW). Epoetin alfa dosing will occur on dialysis days in each Cohort A. Dose adjustment will be per local standard of care (exclusive of IV iron) for routine maintenance of stable Hb levels on dialysis participants.
  Interventions: Drug: Epoetin Alfa
- Cohort B-1 (Roxadustat 1.5 mg/kg TIW) (Experimental): Hyporesponsive participants (with baseline epoetin alfa dosage 125-400 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 1.5 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort B-2 (Roxadustat 2.0 mg/kg TIW) (Experimental): Hyporesponsive participants (with baseline epoetin alfa dosage >115 IU/kg/dose at study entry) will receive roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 6 weeks. Participants who have not completed 6-week treatment at the time of Amendment 2, will continue treatment for up to 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) will be based upon regular monitoring of Hb.
  Interventions: Drug: Roxadustat
- Cohort B (Epoetin Alfa) (Active Comparator): Hyporesponsive participants will receive IV epoetin alfa treatments on Day 1, at their prestudy dose and according to their prestudy dosing schedule (TIW). Epoetin alfa dosing will occur on dialysis days in each Cohort B. Dose adjustment will be per local standard of care (exclusive of IV iron) for routine maintenance of stable Hb levels on dialysis participants.
  Interventions: Drug: Epoetin Alfa
- Cohort B (Placebo) (Placebo Comparator): Hyporesponsive participants will receive placebo matched to roxadustat, administered orally TIW for 19 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be administered per dose and schedule specified in the arms.
  Other Names: FG-4592
  Arms: Cohort A-1 (Roxadustat 1.0 mg/kg TIW); Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg); Cohort A-2 (Roxadustat 1.5 mg/kg TIW); Cohort A-3 (Roxadustat 2.0 mg/kg TIW); Cohort A-4 (Roxadustat 1.8 mg/kg TIW); Cohort A-5 (Roxadustat 1.8 mg/kg TIW); Cohort A-6 (Roxadustat 1.3 mg/kg TIW); Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg); Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg); Cohort A-9 (Roxadustat 2.0 mg/kg); Cohort B-1 (Roxadustat 1.5 mg/kg TIW); Cohort B-2 (Roxadustat 2.0 mg/kg TIW)
Drug: Epoetin Alfa — Epoetin Alfa will be administered per dose and schedule specified in the arms.
  Arms: Cohort B (Epoetin Alfa); Cohorts A (Epoetin Alfa)
Other: Placebo — Placebo matching to roxadustat will be administered per schedule specified in the arm.
  Arms: Cohort B (Placebo)

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of roxadustat in participants with end-stage renal disease (ESRD) on maintenance hemodialysis (HD) therapy, previously treated with intravenous (IV) epoetin alfa.

DETAILED DESCRIPTION:
Dose ranging study with consecutive cohorts in two participant populations: participants normally responding to current anemia treatment (epoetin alfa) ("normoresponders": participants with baseline epoetin alfa dose at study entry 75 to 450 international units [IU]/kilograms [kg]/week) and participants not responding well to current treatment ("hyporesponders": participants with maintenance epoetin alfa dose above 450 IU/kg/week). Normoresponders are randomized to study drug roxadustat or epoetin alfa at a ratio of 3:1; hyporesponders are randomized to study drug roxadustat or epoetin alfa or placebo at a ratio of 2:1:1. The study objectives are to demonstrate that roxadustat is effective in maintaining hemoglobin (Hb) levels when converting from epoetin alfa and to establish optimum starting doses and dose adjustment regimens for Hb maintenance.

ELIGIBILITY:
Key Inclusion Criteria:

* ESRD and receiving maintenance HD TIW for ≥4 months prior to Day 1
* Two most recent Hb values obtained during screening period must be within the ranges set below:

  i) Group A. Normoresponder Criteria: Hb range in the 8 weeks prior to randomization within 9.0 to 13.5 g/dL ii) Group B. Hyporesponder Criteria: Hb range in the 8 weeks prior to randomization within 8.5 to 13.5 g/dL
* Epoetin alfa, dose requirements:

  i) Group A. Normoresponder Criteria - Cohorts A-1 to A-12: Stable IV epoetin alfa dose at baseline (that is, no more than a 30% fluctuation in the weekly dose) during the 4 weeks prior to study Day -3
  1. Cohorts A-1 to A-4: Current and previous (past 4 weeks) epoetin alfa dose range 25 to 85 IU/kg/dose, TIW; weekly dose between 75 and 255 IU/kg/week
  2. Cohort A-5: Current and previous (past 4 weeks) epoetin alfa dose range ≥85 to 115 IU/kg/dose, TIW; total weekly dose between 255 and 450 IU/kg/week
  3. Cohort A-9: Current and previous (past 4 weeks) epoetin alfa dose range ≥85 to 150 IU/kg/dose, TIW; total weekly dose between 255 and 450 IU/kg/week
  4. Cohorts A-6 to A-8: Current and previous (past 4 weeks) epoetin alfa dose range 25 to 115 IU/kg/dose, TIW, and two times a week (BIW); total weekly dose between 75 and 345 IU/kg/week
  5. Cohorts A-10 to A-12: Optional cohorts to be decided (TBD), dosing frequency and dose range to be determined by sponsor ii) Group B. Hyporesponder Criteria:

  <!-- -->

  1. Cohort B-1 (completed): Current and previous (past 4 weeks) epoetin alfa dose range 125 to 400 IU/kg/dose, TIW; weekly dose between 375 and 1200 IU/kg/week
  2. Cohort B-2 to B-4: Current and previous (past 4 weeks) epoetin alfa dose range >115 IU/kg/dose, TIW; total weekly dose >345 IU/kg/week no requirement for stability of epoetin alfa doses
* Complete Blood Count (CBC), Hematology, liver function blood tests, serum folate and vitamin B12 within acceptable limits
* Absence of active or chronic gastrointestinal bleeding
* High sensitivity C-reactive protein (hsCRP) <60 mg/liter for normoresponders Cohorts A-8 through A-12 enrolled under Amendment 3; no hsCRP criteria for hyporesponders
* Body weight: 40 to 140 kg (dry weight)
* Body mass index (BMI): 18 to 45 kg/meter square (m^2)
* Dialysis vascular access via native arteriovenous fistula or synthetic graft, or permanent (tunneled) catheter (not via temporary catheter); permanent and temporary catheters, however, are still prohibited in Cohort A-5

Key Exclusion Criteria:

* Anticipated change in HD prescription
* Any clinically significant infection or evidence of an underlying infection
* Positive for any of the following: Human immunodeficiency virus (HIV); hepatitis B surface antigen (HBsAg); or anti-hepatitis C virus antibody (anti-HCV Ab)
* History of chronic liver disease
* New York Heart Association Class III or IV congestive heart failure
* Chronic inflammatory disease that could impact erythropoiesis (for example, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
* History of myelodysplastic syndrome
* History of hemosiderosis, hemochromatosis, polycystic kidney disease, or anephric
* Active hemolysis or diagnosis of hemolytic syndrome
* Known bone marrow fibrosis
* Uncontrolled or symptomatic secondary hyperparathyroidism
* Any prior organ transplantation
* Drug-treated gastroparesis or short-bowel syndrome
* History of alcohol or drug abuse; or a positive drug screen for a substance that has not been prescribed for the participant
* Prior treatment with roxadustat
* Diagnosis or suspicion of renal cell carcinoma
* Red blood cell (RBC) transfusion within 12 weeks prior to Day 1, or anticipated need for RBC transfusion during the dosing period
* IV iron supplement within 2 weeks prior to Day 1 and/or unwilling to withhold IV iron during the dosing/treatment period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2012-10-15 (Actual); Study Completion 2012-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Franco, Study Director — Kyntra Bio
Locations (25):
- United States (25):
  - Tempe, Arizona
  - Pine Bluff, Arkansas
  - Azusa, California
  - Los Angeles, California
  - Northridge, California
  - Ontario, California
  - Paramount, California
  - Yuba City, California
  - Miami, Florida
  - Pembroke Pines, Florida
  - Honolulu, Hawaii
  - Louisville, Kentucky
  - Detroit, Michigan
  - Kansas City, Missouri
  - Paterson, New Jersey
  - New York, New York
  - Rosedale, New York
  - Williamsville, New York
  - Toledo, Ohio
  - Orangeburg, South Carolina
  - Arlington, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Normoresponder participants were enrolled sequentially in 10 cohorts (A-1 to A-10) with the exception of Cohort A-5 in parallel enrollment with A-6 to A-8. Hyporesponder participants were enrolled in 2 cohorts (B-1 and B-2). Normoresponder participants were those with stable baseline epoetin alfa doses between 75 and 450 international units (IU)/kilogram (kg)/week, while hyporeponders required maintenance epoetin alfa dose above 450 IU/kg/week.
Groups:
- Cohort A-1 (Roxadustat 1.0 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.0 milligrams (mg)/kg, administered orally 3 times weekly (TIW) in the morning of the day after dialysis (interdialytic days) for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target hemoglobin (Hb) values (11.0-13.0 grams [g]/deciliter [dL]) was based upon regular monitoring of Hb.
- Cohort A-2 (Roxadustat 1.5 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.5 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-3 (Roxadustat 2.0 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) received roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-4 (Roxadustat 1.8 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.8 mg/kg, administered orally TIW for 6 weeks. Participants who had not completed 6-week treatment at the time of Amendment 2, continued treatment for up to 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-5 (Roxadustat 1.8 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 85-115 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.8 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-6 (Roxadustat 1.3 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.3 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.3 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 100 mg, and 150 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg); Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.5 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 120 mg, and 200 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-9 (Roxadustat 2.0 mg/kg): Normoresponsive participants (with baseline epoetin alfa dosage 85-150 IU/kg/dose at study entry) received roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohorts A (Epoetin Alfa): Normoresponsive participants received intravenous (IV) epoetin alfa treatments on Day 1, at their prestudy dose and according to their prestudy dosing schedule (TIW). Epoetin alfa dosing occurred on dialysis days in each Cohort A. Dose adjustment was per local standard of care (exclusive of IV iron) for routine maintenance of stable Hb levels on dialysis participants.
- Cohort B-1 (Roxadustat 1.5 mg/kg TIW): Hyporesponsive participants (with baseline epoetin alfa dosage 125-400 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.5 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort B-2 (Roxadustat 2.0 mg/kg TIW): Hyporesponsive participants (with baseline epoetin alfa dosage >115 IU/kg/dose at study entry) received roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 6 weeks. Participants who had not completed 6-week treatment at the time of Amendment 2, continued treatment for up to 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort B (Epoetin Alfa): Hyporesponsive participants received IV epoetin alfa treatments on Day 1, at their prestudy dose and according to their prestudy dosing schedule (TIW). Epoetin alfa dosing occurred on dialysis days in each Cohort B. Dose adjustment was per local standard of care (exclusive of IV iron) for routine maintenance of stable Hb levels on dialysis participants.
- Cohort B (Placebo): Hyporesponsive participants received placebo matched to roxadustat, administered orally TIW for 19 weeks.
Period: Dosing Period 1: 6-Week Treatment
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 2 | 10 | 36 | 4 | 5 | 4 | 4
Received at Least 1 Dose of Study Drug | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 2 | 10 | 36 | 4 | 5 | 4 | 4
Efficacy Evaluable (EE) Population (Received study drug for at least 4 weeks with corresponding Hb measurements or permanently discontinued study medication during the dosing period due to lack of efficacy.) | 9 | 10 | 9 | 11 | 11 | 11 | 11 | 10 | 2 | 10 | 31 | 1 | 3 | 4 | 3
Completed | 10 | 10 | 11 | 10 | 7 | 9 | 9 | 9 | 2 | 8 | 33 | 2 | 1 | 3 | 0
Not Completed | 2 | 2 | 1 | 2 | 5 | 3 | 3 | 3 | 0 | 2 | 3 | 2 | 4 | 1 | 4
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 3 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Other than specified | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Period: Dosing Period 2: 19-Week Treatment
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Started | 0 | 0 | 0 | 7 | 12 | 12 | 12 | 12 | 2 | 10 | 23 | 0 | 5 | 3 | 3
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 7 | 12 | 12 | 12 | 12 | 2 | 10 | 23 | 0 | 5 | 3 | 3
EE Population for 19-week Treatment (Participants randomized designated to receive 19 weeks of study medication and had received study drug for at least 4 weeks with corresponding Hb measurements or permanently discontinued study medication during the dosing period due to lack of efficacy.) | 0 | 0 | 0 | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22 | 0 | 3 | 3 | 2
Completed | 0 | 0 | 0 | 5 | 7 | 9 | 9 | 9 | 2 | 8 | 21 | 0 | 1 | 2 | 0
Not Completed | 0 | 0 | 0 | 2 | 5 | 3 | 3 | 3 | 0 | 2 | 2 | 0 | 4 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Other than specified | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized and received at least 1 dose of study medication.
Groups:
- Cohort A-1 (Roxadustat 1.0 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.0 mg/kg, administered orally TIW in the morning of the day after dialysis (interdialytic days) for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohorts A (Epoetin Alfa): Normoresponsive participants received IV epoetin alfa treatments on Day 1, at their prestudy dose and according to their prestudy dosing schedule (TIW). Epoetin alfa dosing occurred on dialysis days in each Cohort A. Dose adjustment was per local standard of care (exclusive of IV iron) for routine maintenance of stable Hb levels on dialysis participants.
- Total: Total of all reporting groups
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 2 | 10 | 36 | 4 | 5 | 4 | 4 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.1) | 58.8 (13.6) | 56.6 (10.8) | 50.8 (19.4) | 55.2 (10.6) | 58.7 (10.1) | 61.9 (11.9) | 55.7 (14.5) | 57.0 (17.0) | 55.8 (6.8) | 57.9 (11.0) | 55.0 (8.8) | 60.2 (5.9) | 47.0 (12.5) | 58.8 (8.6) | 56.3 (3.680644)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 7 | 5 | 4 | 2 | 5 | 4 | 1 | 3 | 13 | 3 | 5 | 2 | 2 | 61
  Male | 8 | 11 | 5 | 7 | 8 | 10 | 7 | 8 | 1 | 7 | 23 | 1 | 0 | 2 | 2 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Week 7 Hb ≥ Baseline Hb - 0.5 g/dL, Among Normoresponder Participants Treated for 6 Weeks Only
Description: Baseline was defined as the mean of the last 3 Hb values obtained prior to the first dose of study treatment, including Day 1 predose. Last observation carried forward (LOCF) method was used to impute missing values.
Time Frame: Week 7
Population: EE population included participants who received treatment for at least 4 weeks with corresponding Hb measurements not resulted from any rescue therapies including inadvertent use of rescue medication (erythropoiesis-stimulating agent [ESA], IV Iron or red blood cell [RBC] transfusion) or who permanently discontinued study drug during dosing period due to lack of efficacy. Here, 'Overall number of participants analyzed' signifies normoresponder participants who were treated for 6 weeks only.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A-4 (Roxadustat 1.8 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-85 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.8 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A (Epoetin Alfa): Normoresponsive participants received IV epoetin alfa treatments on Day 1, at their prestudy dose and according to their prestudy dosing schedule (TIW). Epoetin alfa dosing occurred on dialysis days in each Cohort A. Dose adjustment was per local standard of care (exclusive of IV iron) for routine maintenance of stable Hb levels on dialysis participants.
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A (Epoetin Alfa)
Number analyzed (Participants) | 9 | 10 | 9 | 5 | 9
Participants | 4 | 8 | 7 | 4 | 3
Statistical Analysis 1: Comparison: Cohort A-1 (Roxadustat 1.0 mg/kg TIW) vs Cohort A (Epoetin Alfa); Test type: Other; p = 1.0000, Fisher Exact — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Cohort A-2 (Roxadustat 1.5 mg/kg TIW) vs Cohort A (Epoetin Alfa); Test type: Other; p = 0.0698, Fisher Exact — Threshold for significance at 0.05 level
Statistical Analysis 3: Comparison: Cohort A-3 (Roxadustat 2.0 mg/kg TIW) vs Cohort A (Epoetin Alfa); Test type: Other; p = 0.1534, Fisher Exact — Threshold for significance at 0.05 level
Statistical Analysis 4: Comparison: Cohort A-4 (Roxadustat 1.8 mg/kg TIW) vs Cohort A (Epoetin Alfa); Test type: Other; p = 0.2657, Fisher Exact — Threshold for significance at 0.05 level

2. Primary Outcome: Number of Participants With Week 7 Hb ≥ Baseline Hb - 0.5 g/dL, Among Hyporesponsive Participants Treated for at Least 6 Weeks
Description: Baseline was defined as the mean of the last 3 Hb values obtained prior to the first dose of study treatment, including Day 1 predose. LOCF method was used to impute missing values.
Time Frame: Week 7
Population: EE population included participants who received treatment for at least 4 weeks with corresponding Hb measurements not resulted from any rescue therapies including inadvertent use of rescue medication (ESA, IV Iron or RBC transfusion) or who permanently discontinued study drug during dosing period due to lack of efficacy.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B-2 (Roxadustat 2.0 mg/kg TIW): Hyporesponsive participants (with baseline epoetin alfa dosage >115 IU/kg/dose at study entry) received roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort B (Placebo): Hyporesponsive participants received placebo matched to roxadustat, administered orally TIW for 6 weeks.
Arm/Group | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 1 | 3 | 4 | 3
Participants | 0 | 1 | 2 | 0
Statistical Analysis 1: Comparison: Cohort B-2 (Roxadustat 2.0 mg/kg TIW) vs Cohort B (Placebo); Test type: Other; p = 1.0000, Fisher Exact — Threshold for significance at 0.05 level

3. Primary Outcome: Number of Participants With a Mean Hb Above 11 g/dL When the Mean Hb Values at Weeks 17, 18, 19, and 20 Were Averaged, Among Participants Treated for 19 Weeks
Description: The average of the mean Hb values that were above 11 g/dL at Weeks 17, 18, 19, and 20 are presented. LOCF method was used to impute missing values.
Time Frame: Weeks 17, 18, 19, and 20
Population: EE population for 19 weeks treatment included all participants randomized designated to receive 19 weeks of study medication and had received study treatment for at least 4 weeks with corresponding Hb measurements not resulted from any rescue therapies including inadvertent use of rescue medication (ESA, IV Iron or RBC transfusion), or who permanently discontinued study medication during the dosing period due to lack of efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22 | 3 | 3 | 2
Participants | 4 | 4 | 6 | 5 | 6 | 2 | 4 | 8 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With a Mean of Hb Within 11-13 g/dL (Values Obtained at Weeks 17, 18, 19, and 20 for Participants Dosed for 19 Weeks)
Description: The average of the mean Hb values that were within 11-13 g/dL at Weeks 17, 18, 19, and 20 are presented. LOCF method was used to impute missing values.
Time Frame: Weeks 17, 18, 19, and 20
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22 | 3 | 3 | 2
Participants | 4 | 1 | 6 | 5 | 6 | 2 | 3 | 8 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With a Mean of Hb Within 10-13 g/dL (Values Obtained at Weeks 17, 18, 19, and 20 for Participants Dosed for 19 Weeks)
Description: The average of the mean Hb values that were within 10-13 g/dL at Weeks 17, 18, 19, and 20 are presented. Because of the small number of hyporesponders enrolled into this study, data for this secondary efficacy analysis as planned per protocol was not collected and summarized for hyporesponder participants. LOCF method was used to impute missing values.
Time Frame: Weeks 17, 18, 19, and 20
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa)
Number analyzed (Participants) | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22
Participants | 5 | 2 | 10 | 10 | 7 | 2 | 6 | 19

6. Secondary Outcome: Change From Baseline in Hb at Week 7 for Participants Treated for at Least 6 Weeks
Description: as for outcome 2
Time Frame: Baseline, Week 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Cohort A-5 (Roxadustat 1.8 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 85-115 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.8 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-6 (Roxadustat 1.3 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.3 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.3 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 100 mg, and 150 mg, respectively, administered as oral capsules for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg); Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.5 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 120 mg, and 200 mg, respectively, administered as oral capsules for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-9 (Roxadustat 2.0 mg/kg): Normoresponsive participants (with baseline epoetin alfa dosage 85-150 IU/kg/dose at study entry) received roxadustat capsules at a dose of 2.0 mg/kg, administered orally TIW for 6 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 9 | 10 | 9 | 11 | 11 | 11 | 11 | 10 | 2 | 10 | 31 | 1 | 3 | 4 | 3
g/dL | -0.40 (1.56) | 0.91 (1.59) | 0.71 (1.61) | 0.25 (1.86) | -0.15 (1.36) | -0.18 (1.55) | -0.32 (1.39) | -0.47 (0.94) | -0.00 (2.12) | 0.24 (1.82) | -0.51 (1.31) | -2.63 | -0.89 (0.74) | -0.28 (0.81) | -2.50 (0.23)

7. Secondary Outcome: Change From Baseline in Hb at Weeks 8, 10, 12, 14, 17, 19, and 20 for Participants Treated for 7-19 Weeks
Description: as for outcome 2
Time Frame: Baseline, Weeks 8, 10, 12, 14, 17, 19, and 20
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22 | 3 | 3 | 2
g/dL
  Change at Week 8 | 0.49 (1.31) | 0.08 (1.56) | 0.01 (1.51) | -0.49 (1.49) | -0.29 (1.09) | 0.05 (2.05) | 0.20 (1.85) | -0.21 (1.02) | -0.89 (0.99) | -0.41 (1.52) | -2.37 (0.00)
  Change at Week 10 | 0.56 (1.49) | 0.17 (1.65) | -0.17 (1.32) | -0.56 (1.35) | -0.27 (1.22) | -0.15 (0.07) | 0.26 (2.07) | -0.34 (1.19) | -1.46 (1.41) | 0.19 (1.48) | -2.37 (0.00)
  Change at Week 12 | 0.26 (1.49) | 0.04 (1.57) | -0.10 (1.42) | -0.56 (1.44) | -0.35 (1.17) | -0.15 (0.92) | 0.38 (2.28) | -0.48 (1.20) | -2.02 (1.47) | -0.08 (2.50) | -2.37 (0.00)
  Change at Week 14 | 0.53 (1.55) | -0.03 (1.73) | -0.27 (1.29) | -0.41 (1.44) | -0.24 (1.68) | -0.15 (1.77) | 0.33 (2.37) | -0.50 (1.23) | -2.29 (1.71) | 0.42 (1.83) | -2.37 (0.00)
  Change at Week 17 | -0.09 (0.88) | -0.09 (1.96) | -0.27 (1.07) | -0.48 (1.42) | -0.27 (1.18) | -0.30 (0.85) | 0.02 (2.06) | -0.45 (1.57) | -2.69 (1.61) | 0.16 (2.27) | -2.37 (0.00)
  Change at Week 19 | -0.11 (1.18) | -0.32 (1.84) | -0.28 (1.07) | -0.82 (1.19) | -0.35 (1.20) | 0.05 (0.07) | -0.10 (2.03) | -0.30 (1.43) | -3.02 (1.08) | 0.12 (2.27) | -2.37 (0.00)
  Change at Week 20 | -0.39 (1.16) | -0.55 (1.88) | -0.55 (1.24) | -0.82 (1.27) | -0.33 (1.34) | 0.15 (0.07) | -0.57 (1.68) | -0.36 (1.50) | -2.82 (1.19) | 0.12 (2.14) | -2.47 (0.14)

8. Secondary Outcome: Number of Participants Who Required Dose Adjustments During the Dosing Period for Participants Treated for 6 Weeks Only
Description: Number of participants who required dose increase, dose reduce, dose interruption or dose resume were reported. Because of the small number of hyporesponders enrolled into this study, data for this secondary efficacy analysis as planned per protocol was not collected and summarized for hyporesponder participants.
Time Frame: Baseline up to Week 6
Population: Safety population included all participants who were randomized and received at least one dose of study medication. Here, 'Overall number of participants analyzed' signifies participants who were treated for 6 weeks only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A (Epoetin Alfa)
Number analyzed (Participants) | 12 | 12 | 12 | 5 | 13
Participants
  Dose Increased | 0 | 3 | 0 | 0 | 9
  Dose Reduced | 0 | 0 | 0 | 2 | 6
  Dose Interrupted | 4 | 7 | 4 | 0 | 3
  Dose Resume | 0 | 6 | 4 | 0 | 0

9. Secondary Outcome: Number of Participants Who Required Dose Adjustments During the Dosing Period for Participants Treated for 19 Weeks
Description: as for outcome 8
Time Frame: Baseline up to Week 19
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa)
Number analyzed (Participants) | 7 | 12 | 12 | 12 | 12 | 2 | 10 | 23
Participants
  Dose Increased | 2 | 5 | 5 | 4 | 7 | 1 | 8 | 12
  Dose Reduced | 3 | 3 | 5 | 4 | 4 | 1 | 6 | 11
  Dose Interrupted | 1 | 5 | 2 | 0 | 1 | 0 | 3 | 9
  Dose Resume | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 8

10. Secondary Outcome: Number of Participants Whose Hb Levels Were Maintained at Week 7 to Within ±1 g/dL of Their Mean 4-Week Screening Period Baseline Value for Participants Treated for At Least 6 Weeks
Time Frame: Week 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 9 | 10 | 9 | 11 | 11 | 11 | 11 | 10 | 2 | 10 | 31 | 1 | 3 | 4 | 3
Participants | 3 | 3 | 5 | 5 | 4 | 3 | 6 | 6 | 0 | 1 | 19 | 0 | 2 | 3 | 0

11. Secondary Outcome: Number of Participants Whose Hb Levels Were Maintained at Week 7 to Within ±1 g/dL of Their Mean 4-Week Screening Period Baseline Value for Participants Treated for 19 Weeks
Time Frame: Week 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22 | 3 | 3 | 2
Participants | 3 | 4 | 3 | 6 | 6 | 0 | 1 | 13 | 2 | 3 | 0

12. Secondary Outcome: Number of Participants Treated for 6 Weeks Only Whose Hb Levels at Week 7 Were Greater Than Their Baseline Level
Description: Baseline was defined as the mean of the last 3 Hb values obtained prior to the first dose of study treatment, including Day 1 predose. LOCF method was used to impute missing values. Because of the small number of hyporesponders enrolled into this study, data for this secondary efficacy analysis as planned per protocol was not collected and summarized for hyporesponder participants.
Time Frame: Week 7
Population: EE population included participants who received treatment for at least 4 weeks with corresponding Hb measurements not resulted from any rescue therapies including inadvertent use of rescue medication (ESA, IV Iron or RBC transfusion) or who permanently discontinued study drug during dosing period due to lack of efficacy. Here, 'Overall number of participants analyzed' signifies participants who were treated for 6 weeks only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A (Epoetin Alfa)
Number analyzed (Participants) | 9 | 10 | 9 | 5 | 9
Participants | 3 | 7 | 6 | 3 | 2

13. Secondary Outcome: Number of Participants Treated for 7-19 Weeks Whose Hb Levels at Weeks 8, 10, 12, 14, 17, 19, and 20 Were Greater Than Their Baseline Level
Description: as for outcome 12
Time Frame: Weeks 8, 10, 12, 14, 17, 19, and 20
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A-6 (Roxadustat 1.3 mg/kg TIW): Normoresponsive participants (with baseline epoetin alfa dosage 25-125 IU/kg/dose at study entry) received roxadustat capsules at a dose of 1.3 mg/kg, administered orally TIW for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-125 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.3 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 100 mg, and 150 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
- Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-125 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.5 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 120 mg, and 200 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring of Hb.
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa)
Number analyzed (Participants) | 6 | 11 | 11 | 11 | 10 | 2 | 10 | 22
Participants
  Week 8 | 3 | 6 | 4 | 4 | 4 | 1 | 6 | 9
  Week 10 | 3 | 6 | 4 | 4 | 5 | 0 | 6 | 7
  Week 12 | 3 | 6 | 6 | 4 | 3 | 1 | 5 | 9
  Week 14 | 3 | 6 | 6 | 4 | 1 | 1 | 6 | 6
  Week 17 | 2 | 5 | 5 | 4 | 4 | 1 | 6 | 6
  Week 19 | 2 | 4 | 5 | 2 | 4 | 1 | 6 | 8
  Week 20 | 3 | 3 | 5 | 2 | 5 | 2 | 5 | 7

14. Secondary Outcome: Number of Participants Who Required Rescue Anemia Treatment Due to Hb Levels, Among Participants Treated for at Least 6 Weeks
Description: Rescue anemia treatment included any ESA dosing, RBC transfusion, or IV iron.
Time Frame: Baseline up to Week 6
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 2 | 10 | 36 | 4 | 5 | 4 | 4
Participants | 2 | 2 | 3 | 4 | 2 | 3 | 2 | 3 | 0 | 4 | 6 | 1 | 3 | 0 | 1

15. Secondary Outcome: Number of Participants Who Required Rescue Anemia Treatment Due to Hb Levels, Among Participants Treated for 19-Weeks
Description: Rescue anemia treatment included any ESA dosing, RBC transfusion, or IV iron.
Time Frame: Baseline up to Week 19
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 7 | 12 | 12 | 12 | 12 | 2 | 10 | 23 | 5 | 3 | 3
Participants | 4 | 2 | 3 | 2 | 3 | 0 | 4 | 4 | 3 | 0 | 1

16. Secondary Outcome: Number of Participants Requiring Dose Reduction Secondary to Excessive Erythropoiesis During Dosing Period, Among Participants Treated for at Least 6-Weeks
Time Frame: Baseline up to Week 6
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg): Normoresponsive participants (with baseline epoetin alfa dosage 25-115 IU/kg/dose at study entry) received tiered, weight-based initial doses of roxadustat (approximately 1.3 mg/kg/dose TIW). Low weight (40 to 60 kg), medium weight (>60 to 90 kg), and heavy weight (>90 to 140 kg) participants received roxadustat 70 mg, 100 mg, and 150 mg, respectively, administered as oral capsules for 19 weeks. Dose adjustment to achieve correction and subsequent maintenance of target Hb values (11.0-13.0 g/dL) was based upon regular monitoring o
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 2 | 10 | 36 | 4 | 5 | 4 | 4
Participants | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 4 | 6 | 0 | 0 | 1 | 0

17. Secondary Outcome: Number of Participants Requiring Dose Reduction Secondary to Excessive Erythropoiesis During Dosing Period, Among Participants Treated for 19-Weeks
Time Frame: Baseline up to Week 19
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 7 | 12 | 12 | 12 | 12 | 2 | 10 | 23 | 5 | 3 | 3
Participants | 0 | 0 | 2 | 1 | 2 | 1 | 4 | 6 | 0 | 1 | 0

18. Secondary Outcome: Rate of Change in Hb Levels, Measured by Regression Slopes of the Hb Values During Treatment up to Week 6
Description: The rate of rise was computed as the slope of the regression line of change in Hb level (in g/dL) vs. time (in weeks) using Random Coefficient Model. Because of the small number of hyporesponders enrolled into this study, data for this secondary efficacy analysis as planned per protocol was not collected and summarized for hyporesponder participants.
Time Frame: Baseline up to Week 6
Population: EE included participants who received treatment for at least 4 weeks with corresponding Hb measurements not resulted from any rescue therapies including inadvertent use of rescue medication (ESA, IV Iron or RBC transfusion) or who permanently discontinued study drug during dosing period due to lack of efficacy. Here, 'Overall number of participants analyzed' signifies participants who were treated for 6 weeks only.
Measure: Number; unit: g/dL/week
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A (Epoetin Alfa)
Number analyzed (Participants) | 9 | 10 | 9 | 5 | 9
g/dL/week | -0.0135 | 0.1926 | 0.1682 | -0.0220 | -0.1267

19. Secondary Outcome: Trough Plasma Concentration of Roxadustat and Epoetin Alfa
Time Frame: Predose, 4, 8, 12, 24, 48, and 72 hours postdose at Weeks 1 and 6
Population: Data for trough plasma concentration of roxadustat and epoetin alfa were not collected for this study.
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 23
Description: Safety population included all participants who were randomized and received at least one dose of study medication.
Arm/Group | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) | Cohort A-9 (Roxadustat 2.0 mg/kg) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) | Cohorts A (Epoetin Alfa) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) | Cohort B (Epoetin Alfa) | Cohort B (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/12 | 3/12 | 0/12 | 4/12 | 5/12 | 3/12 | 5/12 | 3/12 | 0/2 | 3/10 | 6/36 | 2/4 | 2/5 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/12 | 1/12 | 1/12 | 4/12 | 2/12 | 2/12 | 1/12 | 2/12 | 0/2 | 3/10 | 2/36 | 3/4 | 2/5 | 0/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) (N=12) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) (N=12) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) (N=12) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) (N=12) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) (N=12) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) (N=12) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) (N=12) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) (N=12) | Cohort A-9 (Roxadustat 2.0 mg/kg) (N=2) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) (N=10) | Cohorts A (Epoetin Alfa) (N=36) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) (N=4) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) (N=5) | Cohort B (Epoetin Alfa) (N=4) | Cohort B (Placebo) (N=4)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A-1 (Roxadustat 1.0 mg/kg TIW) (N=12) | Cohort A-2 (Roxadustat 1.5 mg/kg TIW) (N=12) | Cohort A-3 (Roxadustat 2.0 mg/kg TIW) (N=12) | Cohort A-4 (Roxadustat 1.8 mg/kg TIW) (N=12) | Cohort A-5 (Roxadustat 1.8 mg/kg TIW) (N=12) | Cohort A-6 (Roxadustat 1.3 mg/kg TIW) (N=12) | Cohort A-7 (Weight Tiered Roxadustat 70-100-150 mg) (N=12) | Cohort A-8 (Weight Tiered Roxadustat 70-120-200 mg) (N=12) | Cohort A-9 (Roxadustat 2.0 mg/kg) (N=2) | Cohort A-10 (Weight Tiered Roxadustat 70-120-200 mg) (N=10) | Cohorts A (Epoetin Alfa) (N=36) | Cohort B-1 (Roxadustat 1.5 mg/kg TIW) (N=4) | Cohort B-2 (Roxadustat 2.0 mg/kg TIW) (N=5) | Cohort B (Epoetin Alfa) (N=4) | Cohort B (Placebo) (N=4)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes